CLINICAL TRIAL: NCT06099236
Title: A Prospective, Non-interventional, Observational Study of Presentation, Treatment Patterns and Outcomes in Chinese Atypical Hemolytic Uremic Syndrome Patients
Brief Title: A Prospective, Non-interventional, Observational Study of Presentation, Treatment Patterns and Outcomes in Atypical Hemolytic Uremic Syndrome Patients
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D7413R00001
Record Dates: First submitted 2023-09-29; First posted 2023-10-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Atypical Hemolytic Uremic Syndrome(aHUS)
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
This is a China, non-interventional, observational study and will follow the Good Phar-macoepidemiology Practices guidelines.

This study will enrol paediatric and adult patients diagnosed with aHUS who will be treated according to routine clinical practice defined by local institutional treatment guidelines/protocol. Those aHUS patients who will be treated with a supportive therapy, which does not contain eculizumab, will be monitored for up to 12 months since the ini-tial diagnosis. Patients initiated on eculizumab treatment anytime between aHUS diagno-sis until 12 months will be followed for additional 12 months, starting from the ecu initia-tion. Patient disposition, characteristics, outcomes and safety will be described for all pa-tients enrolled into this study

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study. Age

1. Patients of any age, who are diagnosed as aHUS by a professional physician (first epi-sode or relapse).

   Type of Patient and Disease Characteristics
2. Evidence of TMA, including thrombocytopenia, evidence of hemolysis, and kidney dys-function, based on the following laboratory findings, should be recorded within 2 weeks time frame:

   1. Platelet count < 150,000 per microliter (μL), and
   2. Mechanic hemolytic anemia evident by LDH ≥ 1.5 × upper limit of normal (ULN), and hemoglobin ≤ lower limit of normal (LLN) for age and gender and
   3. Serum creatinine level ≥ ULN in adults (≥18 years of age), or ≥ 97.5th percentile for age at screening in children (patients who require dialysis for acute kidney injury are also eligi-ble).
3. Gender: Male and/or female. Informed Consent
4. Willing and able to give written informed consent and comply with the study visit schedule as described in Section 6.2.1. For patients < 18 years of age, patient's legal guardian must be willing and able to give written informed consent and the patient must be willing to give written informed assent (if applicable as determined by the central.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions

1. Patients who were diagnosed with HUS only due to Shiga toxin-producing Escherichia coli (STEC).
2. Patients who were diagnosed with TTP (ADAMTS13 activity <10%). Other Exclusions
3. Unable to give written informed consent.
4. Any medical or psychological condition that, in the opinion of the Investigator, could increase the risk to the participant by participating in the study or confound the outcome of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: paediatric and adult patients diagnosed with aHUS
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Event free survival, where event defined as ESRD or death on or after TMA onset. | 12 Months

SECONDARY OUTCOMES:
Death | 12 Months
End-stage renal disease(ESRD) | 12 Months
Complete TMA Response during observation the as evidenced by simultaneous normalization of hemato-logical parameters (platelet count and LDH) and ≥ 25% improvement in serum creatinine from baseline | 12 Months
Complete Thrombotic Microangiopathy(TMA ) Response status over time | 12 Months
Time to Complete Thrombotic Microangiopathy(TMA ) Response | 12 Months
Thrombotic Microangiopathy(TMA ) relapse | 12 Months
Observed value and change from baseline in estimated glomerular filtration rate (eGFR) | 12 Months
Chronic kidney disease (CKD) stage, as evaluated by the Investigator and classified as improved, stable (no change), or worsened compared to baseline | 12 Months
Proteinuria over time. | 12 Months
Urine protein-to-creatinine ratio over time. | 12 Months
Plasma C3, C4, CH50, Factor H and I, soluble C5b-9 (sC5b-9) and CD46 expression over time. | 12 Months
The proportion of patients with normal platelet count (≥150 x 109/L),LDH levels ≤upper limit of normal , serum creatinine < up-per limit of normal for age or an improvement > 25% compared to baseline,eGFR≥ 60 mL/min/1.73 m2, proteinuria negative. | 12 Months
Descriptive data of events of interest (serious infec-tions (Aspergillus infections and infections due to en-capsulated bacteria such as Neisseria meningitidis), pregnancy, lactation, and follow-up-data on neonates for 3 months after delivery) | 12 Months
Descriptive data of Serious Adverse Events (SAEs) for treatment period 2. | 12 Months
Observed Value in Platelet Count | 12 Months
Observed Value in Lactate Dehydrogenase (LDH) (mg/dL) | 12 Months
Observed Value in Hemoglobin (mg/dL) | 12 Months
Change from Baseline in Platelet Count | 12 Months
Change from Baseline in Lactate Dehydrogenase (LDH) (mg/dL) | 12 Months
Change from Baseline in Hemoglobin (mg/dL) | 12 Months
The number of patients still on dialysis during each follow-up visit | 12 Months

CONTACTS AND LOCATIONS:
Locations (26):
- China (26):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Chongqing, Sichuan
  - Research Site, Anhui
  - Research Site, Beijing
  - Research Site, Chongqing
  - Research Site, Fujian
  - Research Site, Guangdong
  - Research Site, Guangxi
  - Research Site, Guizhou
  - Research Site, Hainan
  - Research Site, Hebei
  - Research Site, Henan
  - Research Site, Hong Kong
  - Research Site, Hubei
  - Research Site, Hunan
  - Research Site, Jiangsu
  - Research Site, Jiangxi
  - Research Site, Liaoning
  - Research Site, Shaanxi
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shanxi
  - Research Site, Sichuan
  - Research Site, Tianjin
  - Research Site, Xinjiang
  - Research Site, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/